CLINICAL TRIAL: NCT05428579
Title: Status of Surgical Resection and Histologic Subtype as Predictors of Local Recurrence in Retroperitoneal Liposarcoma - Case Series
Brief Title: Status of Surgical Resection and Histologic Subtype as Predictors of Local Recurrence in Retroperitoneal Liposarcoma
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Edivaldo Massazo Utiyama, Full Professor of III General Surgery Division, University of Sao Paulo General Hospital
Other Study IDs: 29071984
Record Dates: First submitted 2019-04-09; First posted 2022-06-23 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Liposarcoma of Soft Tissue; Surgical Procedure, Unspecified
Keywords: retroperitoneal liposarcoma; overall survival; local recurrence free survival
MeSH Terms: conditions — Retroperitoneal liposarcoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Retroperitoneal Liposarcoma resection — Retroperitoneal Liposarcoma resection

SUMMARY:
Soft tissue sarcomas are rare malignant tumors. Liposarcoma constitute the most frequent histological subtype of retroperitoneal sarcoma. The prognosis of soft tissue sarcomas depend on clinical and histologic characteristics. Objective: Evaluate variables that may be related to overall survival and local recurrence free survival in patients with retroperitoneal liposarcoma. Methods: retrospective analysis of medical records of 60 patients attended from 1997 to 2017, who underwent surgical resection of retroperitoneal liposarcoma.

ELIGIBILITY:
Inclusion Criteria:

* All patients who underwent surgical resection of retroperitoneal liposarcoma

Exclusion Criteria:

* Unresectable disease (upper mesenteric artery or vein involvement) or metastatic disease (sarcomatosis or distant disease)

Ages: 17 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 60 patients attended at the University of São Paulo Medical School Hospital (HC-FMUSP) and the Cancer Institute of the State of São Paulo (ICESP) from 1997 to 2017, who underwent surgical resection of the primary tumor at these institutions, as well as those referred after resection at other services.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Overall survival rate | 60 months
Local recurrence-free survival rate | 60 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Neuhaus SJ, Barry P, Clark MA, Hayes AJ, Fisher C, Thomas JM. Surgical management of primary and recurrent retroperitoneal liposarcoma. Br J Surg. 2005 Feb;92(2):246-52. doi: 10.1002/bjs.4802. PMID 15505870
- [Result] Singer S, Antonescu CR, Riedel E, Brennan MF. Histologic subtype and margin of resection predict pattern of recurrence and survival for retroperitoneal liposarcoma. Ann Surg. 2003 Sep;238(3):358-70; discussion 370-1. doi: 10.1097/01.sla.0000086542.11899.38. PMID 14501502